CLINICAL TRIAL: NCT00864214
Title: A Pharmacokinetic Evaluation of Bioidentical Compounded Estrogen Cream and Natural Progesterone
Acronym: HRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Richa Sood, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-006363; 08-000223
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Menopause
Keywords: bioidentical hormone; menopause; estrogen; progesterone
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Estrogen is the Biest 2.0 mg bioidentical cream; the placebo is the transdermal patch; the progesterone is compounded progesterone-100 mg
  Interventions: Drug: bioidentical hormone (Biest)
- 2 (Experimental): Estrogen is the Biest 2.5 mg bioidentical cream; the placebo is the transdermal patch; the progesterone is compounded progesterone-100 mg
  Interventions: Drug: bioidentical hormone (Biest)
- 3 (Experimental): Estrogen is the Biest 3.0 mg bioidentical cream; the placebo is the transdermal patch; the progesterone is compounded progesterone-100 mg
  Interventions: Drug: bioidentical hormone (Biest)
- 4 (Experimental): Estrogen is the Vivelle-Dot patch 0.05 mg; the placebo is the transdermal cream; the progesterone is micronized progesterone-100 mg
  Interventions: Drug: bioidentical hormone (Vivelle-Dot)

INTERVENTIONS:
Drug: bioidentical hormone (Biest) — Estrogen is the Biest 2.0 mg bioidentical cream; the placebo is the transdermal patch; the progesterone is compounded progesterone-100 mg
  Arms: 1
Drug: bioidentical hormone (Biest) — Estrogen is the Biest 2.5 mg bioidentical cream; the placebo is the transdermal patch; the progesterone is compounded progesterone-100 mg
  Arms: 2
Drug: bioidentical hormone (Biest) — Estrogen is the Biest 3.0 mg bioidentical cream; the placebo is the transdermal patch; the progesterone is compounded progesterone-100 mg
  Arms: 3
Drug: bioidentical hormone (Vivelle-Dot) — Estrogen is the Vivelle-Dot patch 0.05 mg; the placebo is the transdermal cream; the progesterone is micronized progesterone-100 mg
  Arms: 4

SUMMARY:
Bioidentical compounded hormone therapy (BCHT) is considered a 'safer' option to the conventional hormones (HT) by its proponents. However, there is limited research data to support their claims. Our group at the Women's Health Clinic, in collaboration with the Departments of Endocrinology, Complementary Medicine and Laboratory Medicine, is interested in developing a line of research to test the safety and efficacy of BCHT. In the present study, we aim to find the dose of BCHT that is bioequivalent to conventional HT, in a randomized, blinded, four-arm, phase I clinical trial. We will estimate the levels of estrone (E1), estradiol (E2) and estriol (E3) at baseline and at steady state with two-weeks of administration of three commonly used doses of bioidentical compounded estrogen cream (Biest) and a standard dose conventional estrogen patch (Vivelle-Dot). E1, E2, and E3 values will be summarized using point estimates and 95% confidence intervals. Two-sample t-test will be used to compare each Biest group to the Vivelle-Dot group. Healthy postmenopausal women, with no contraindications for hormone use, who are able to fully understand and participate in the trial, will be enrolled. We will utilize the resources of Mayo CRU to conduct this study.

DETAILED DESCRIPTION:
This study is designed as a Phase I, blinded, randomized, four-arm clinical trial. Participants will be randomized to one of the four interventions: Biest transdermal cream 2.0 mg/0.5 g daily, Biest 2.5 mg/0.5 g daily, Biest 3.0 mg/0.5 g daily or Vivelle-Dot patch 0.05 mg/24 hours changed biweekly. Serum levels of E1, E2, E3 and progesterone will be obtained at baseline before starting the intervention and then multiple times on days 1 15 and 16 of study, as outlined in the table below (Table 3.1). The peak and steady state concentrations of E1, E2 and E3, along with time to reach the peak levels, and area under the curve will be calculated. Baseline and steady state levels of progesterone will also be compared between the compounded and micronized progesterone groups. If there are abnormalities in estrogen levels or symptoms suggesting such, a vaginal ultrasound would be done to exclude possible ovarian activity as a source.

ELIGIBILITY:
Inclusion Criteria:

1. Women 40-60 years old;
2. Postmenopausal status, as documented by absence of periods for ≥ 1 year or amenorrhea for ≥ 6 months along with FSH ≥ 40 IU/L;
3. Surgical menopause;
4. History of a normal mammogram within the last 11 months;
5. Normal screening labs (within 20% of upper limit of lab normal);
6. Able to understand and sign informed consent; and
7. Able and willing to be in a monitored CRU setting and provide blood samples as requested.

Exclusion Criteria:

1. Contraindications to the use of hormones because of personal history of coronary artery disease, stroke, breast cancer, DVT/PE, active liver or gall bladder disease, hormone dependent migraine headaches, endometrial, ovarian or other hormone dependent cancers;
2. Medical conditions increasing the risk of complications from hormone replacement such as uncontrolled hypertension (>160/100 mmHg), smoking, diabetes and lupus;
3. Current use of estrogen, progesterone or testosterone;Depending on the drug, it could be 7 days to 6 months.
4. Current use of isoflavone containing products;
5. Current use of protein binding medications like rifampin, warfarin, antiepileptic drugs (effect on estrogen bioavailability);
6. Family history of premenopausal breast cancer in a first degree relative, two or more premenopausal breast cancers in second degree relatives, male breast cancer, ovarian cancer in two or more relatives and; and
7. Women with alcohol or substance abuse or dementia (compliance issues).
8. Women who are more than ten years from their last menstrual period (unfavorable risk : benefit ratio)
9. Women with peanut allergy (Prometrium has peanut oil)
10. Women who are found to have premenopausal estrogen levels, as confirmed by a baseline Estradiol level of >35 pg/ml and vaginal ultrasound suggesting ovarian activity.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To measure estrone, estradiol and estriol levels at baseline and after achieving a steady state with 15-days of administration of three commonly used doses of bioidentical compounded estrogen cream and a standard dose conventional estrogen patch. | Day 1 and Day 15
To measure the progesterone levels at baseline and after achieving a steady state with 15-days of administration of 100 mg/day of two different oral progesterone formulations. | Day 1 and Day 15

SECONDARY OUTCOMES:
To assess the feasibility of conducting a clinical trial randomizing patients to daily estradiol-estriol transdermal cream or biweekly estradiol patch for 15 days in 40 healthy postmenopausal women. | Day 1 and Day 15
To assess the tolerability of use of daily estradiol-estriol transdermal cream and biweekly estradiol patch for 15 days in 40 healthy postmenopausal women in a randomized clinical trial. | Day 1 and Day 15
To test if genetic variation in SULT1A1 copy number and single nucleotide polymorphisms (SNPs) influences estrogen pharmacokinetics in 40 healthy postmenopausal women receiving exogenous estrogen therapy. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Richa Sood, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Sood R, Warndahl RA, Schroeder DR, Singh RJ, Rhodes DJ, Wahner-Roedler D, Bahn RS, Shuster LT. Bioidentical compounded hormones: a pharmacokinetic evaluation in a randomized clinical trial. Maturitas. 2013 Apr;74(4):375-82. doi: 10.1016/j.maturitas.2013.01.010. Epub 2013 Feb 4. PMID 23384975